CLINICAL TRIAL: NCT01675453
Title: The Efficacy and Safety of 7.2% NaCl Plus 6% Hydroxyethyl 200/0.5 in Patients Scheduled for First-time Coronary Artery Bypass Grafting With Cardiopulmonary Bypass.
Brief Title: The Efficacy and Safety of Hypertonic Saline in Cardiac Surgery Patients.
Acronym: ESHHS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Evgeny Fominskiy, MD, PhD, Anesthesiologist, Meshalkin Research Institute of Pathology of Circulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ESHHS
Record Dates: First submitted 2012-08-05; First posted 2012-08-30 (Estimated); Results first posted 2014-06-19 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-04

CONDITIONS: Coronary Artery Disease; Edema
Keywords: Organ dysfunction; Hypertonic solution; Extravascular water; Cardiopulmonary Bypass
MeSH Terms: conditions — Coronary Artery Disease; Edema | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 7.2% NaCl /hydroxyethyl starch 200/0.5 (Active Comparator): On-pump CABG. 7.2% NaCl plus 6% hydroxyethyl starch 200/0.5 solution (HyperHAES) 4 mL/kg for 30 min, IV (in the vein), once, starting after the first hemodynamic measurement is obtained (before the beginning of CPB)
  Interventions: Drug: 7.2% NaCl plus 6% hydroxyethyl starch 200/0.5
- 0.9% NaCl (Placebo Comparator): On-pump CABG. 0.9% NaCl (isotonic saline) 4 mL/kg for 30 min, IV (in the vein), once, starting after the first hemodynamic measurement is obtained (before the beginning of CPB)
  Interventions: Drug: 0.9% NaCl

INTERVENTIONS:
Drug: 7.2% NaCl plus 6% hydroxyethyl starch 200/0.5
  Other Names: HyperHAES
  Arms: 7.2% NaCl /hydroxyethyl starch 200/0.5
Drug: 0.9% NaCl
  Other Names: Saline
  Arms: 0.9% NaCl

SUMMARY:
The organ dysfunction following cardiopulmonary bypass (CPB) occurs frequently in cardiac surgery patients. Systemic inflammatory response initiated by CPB through releasing of several mediators lead to altered endothelial integrity and in consequence the leakage of proteins and fluids from the intravascular to the interstitial compartment is occurred. Increased capillary permeability and decreased colloid osmotic pressure were shown to play a key role for fluid shift and increasing of extravascular water. Further tissue edema can result in injury to many organs, including the heart, lungs, brain, kidneys and can lead to adverse outcomes.

Hypertonic solution creates an osmotic gradient across the cellular membrane, causing a fluid shift from the intracellular and the interstitial spaces of tissue into the intravascular compartment.

The purpose of this study is to investigate the efficacy and safety of 7.2% NaCl plus 6% hydroxyethyl starch 200/0.5 in patients scheduled for first-time coronary artery bypass grafting with cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for first-time coronary artery bypass grafting with cardiopulmonary bypass

Exclusion Criteria:

* age >70 years
* body mass index <18 and >35 kg/m2
* left ventricular ejection fraction <40%
* myocardial infarction <6 months before surgery
* stroke or transient ischemic attack <12 months before surgery
* diabetes mellitus
* glomerular filtration rate <90 mL/min
* emergency surgery
* hematocrit <30%.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir V Lomivorotov, MD, PhD, Principal Investigator — Novosibirsk Research Institute of Pathology of Circulation
Locations (1):
- Novosibirsk Research Institute of Pathology of Circulation, Novosibirsk, Novosibirsk Territory, Russia

REFERENCES:
- [Derived] Lomivorotov VV, Fominskiy EV, Efremov SM, Nepomniashchikh VA, Lomivorotov VN, Chernyavskiy AM, Shilova AN, Karaskov AM. Infusion of 7.2% NaCl/6% hydroxyethyl starch 200/0.5 in on-pump coronary artery bypass surgery patients: a randomized, single-blind pilot study. Shock. 2014 Mar;41(3):193-9. doi: 10.1097/SHK.0000000000000087. PMID 24549094

RESULTS

PARTICIPANT FLOW:
Groups:
- 7.2% NaCl /Hydroxyethyl Starch 200/0.5 (Study Group): On-pump CABG. 7.2% NaCl plus 6% hydroxyethyl starch 200/0.5 solution (HyperHAES) 4 mL/kg for 30 min, IV (in the vein), once, starting after the first hemodynamic measurement is obtained (before the beginning of CPB)
  7.2% NaCl plus 6% hydroxyethyl starch 200/0.5
- 0.9% NaCl (Control Group): On-pump CABG. 0.9% NaCl (isotonic saline) 4 mL/kg for 30 min, IV (in the vein), once, starting after the first hemodynamic measurement is obtained (before the beginning of CPB)
  0.9% NaCl
Period: Overall Study
Arm/Group | 7.2% NaCl /Hydroxyethyl Starch 200/0.5 (Study Group) | 0.9% NaCl (Control Group)
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 7.2% NaCl /Hydroxyethyl Starch 200/0.5 (Study Group) | 0.9% NaCl (Control Group) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [54 to 63] | 57 [51 to 63] | 58 [51 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 15 | 19 | 34
Region of Enrollment [Number; unit: participants]
  Russian Federation | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Extravascular Lung Water Index
Description: Extravascular lung water index (ELWI; mL/kg) will be used to assess this outcome measure. ELWI was monitored by transcardiopulmonary thermodilution technique with the PiCCO plus system. Extravascular lung water represents the extravascular fluid of the lung tissue. It includes intra-cellular, interstitial and intra-alveolar water (not pleural effusion). It is indexed to "Predicted Body Weight".
Time Frame: baseline; 5 min after infusion; 5 min after CPB; 30 min after CPB; end of surgery; 2 h, 4 h, 6 h, 12 h after CPB; Postoperative day 1
Measure: Median (Inter-Quartile Range); unit: mL/kg
Arm/Group | 7.2% NaCl /Hydroxyethyl Starch 200/0.5 (Study Group) | 0.9% NaCl (Control Group)
Number analyzed (Participants) | 20 | 20
mL/kg
  baseline | 9 [8 to 10] | 8 [8 to 9]
  5 min after infusion | 9 [8 to 10] | 8 [8 to 10]
  5 min after CPB | 9 [8 to 9] | 10 [9 to 10]
  30 min after CPB | 9 [8 to 9] | 9 [9 to 10]
  end of surgery | 8 [8 to 9] | 9 [8 to 10]
  2 h after CPB | 8 [8 to 9] | 9 [8 to 10]
  4 h after CPB | 7 [6 to 8] | 9 [8 to 10]
  6 h after CPB | 7 [6 to 7] | 9 [8 to 10]
  12 h after CPB | 7 [6 to 8] | 9 [8 to 10]
  POD 1 | 7 [7 to 8] | 9 [8 to 10]

2. Secondary Outcome: Pulmonary Oxygenation
Description: Index of arterial oxygenation efficiency (PaO2/FiO2), alveolar-arterial oxygen tension difference (AaDO2) will be used to assess this outcome measure.
Time Frame: 24 hours
Reporting Status: Not Posted

3. Secondary Outcome: Oxygen Delivery
Description: Oxygen delivery index (DO2I) will be used to assess this outcome measure.
Time Frame: 24 hours
Reporting Status: Not Posted

4. Secondary Outcome: Cardiac Index
Time Frame: 24 hours
Reporting Status: Not Posted

5. Secondary Outcome: Fluid Balance
Description: Net fluid balance at the end of surgery equals the sum of all infusions minus the urine output. Net fluid balance at postoperative day 1 equals the sum of all infusions minus the urine output and blood loss.
Time Frame: 24 hours
Reporting Status: Not Posted

6. Secondary Outcome: Inflammation Response
Description: Serum levels of Interleukin 6 (IL-6) and Interleukin 10 (IL-10) will be used to assess this outcome measure.
Time Frame: 24 hours
Reporting Status: Not Posted

7. Secondary Outcome: Endothelial Integrity
Description: Serum levels of intercellular adhesion molecule-1 (ICAM-1), E-selectin will be used to assess this outcome measure.
Time Frame: 24 hours
Reporting Status: Not Posted

8. Secondary Outcome: Plasma Na
Time Frame: 24 hours
Reporting Status: Not Posted

9. Secondary Outcome: Plasma Osmolarity
Time Frame: 24 hours
Reporting Status: Not Posted

10. Secondary Outcome: Rate of Acute Kidney Injury
Description: serum creatinine, serum cystatin C, urine neutrophil gelatinase-associated lipocalin (uNGAL) will be used to asses this outcome measure.
Time Frame: 48 hours
Reporting Status: Not Posted

11. Secondary Outcome: Rate of Hyperchloremic Metabolic Acidosis
Description: blood pH, base excess (BE), plasma level of Cl will be used to assess this outcome measure.
Time Frame: 24 hours
Reporting Status: Not Posted

12. Secondary Outcome: Stroke Volume Index
Time Frame: 24 hours
Reporting Status: Not Posted

13. Secondary Outcome: Rate of Neurological Complications
Description: Delirium, clinically diagnosed stroke, and encephalopathy.
Time Frame: 24 hours
Reporting Status: Not Posted

14. Secondary Outcome: Blood Loss
Description: Bleeding from chest tubes
Time Frame: 24 hours
Reporting Status: Not Posted

15. Secondary Outcome: Duration of Mechanical Ventilation
Time Frame: 24 hours
Reporting Status: Not Posted

16. Secondary Outcome: Chloride Loading
Description: The amount of chloride ions (mmol per patient) which will be infused during the surgery and ICU stay
Time Frame: 24 h
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | 7.2% NaCl /Hydroxyethyl Starch 200/0.5 (Study Group) | 0.9% NaCl (Control Group)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes